CLINICAL TRIAL: NCT02174913
Title: Awakening in Spine Surgery Patients Having Neurophysiologic Monitoring: A Comparison Study Between Clinical Signs and Bispectral Index (BIS) Guided Target Controlled Infusion(TCI) of Propofol
Brief Title: Awakening in Spine Surgery: A Comparison Between Clinical Signs and Bispectral Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 099/2557
Record Dates: First submitted 2014-06-12; First posted 2014-06-26 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Spine Diseases
Keywords: Awakening time; Bispectral index; clinical signs; neurophysiologic monitoring; spine surgery
MeSH Terms: conditions — Spinal Diseases; Signs and Symptoms | interventions — Consciousness Monitors; Fentanyl; Atracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bispectral index/TCI propofol/fentanyl (Active Comparator): Bispectral index guides the target controlled infusion of propofol by keeping BIS 40-60 throughout operation. Fentanyl is used for analgesia and atracurium is used for tracheal intubation.
  Interventions: Device: bispectral index; Drug: Target controlled infusion of propofol; Drug: Fentanyl; Drug: Atracurium
- clinical signs/TCI propofol/fentanyl (Placebo Comparator): Clinical signs (heart rate, blood pressure and movement) guide target controlled infusion(TCI) of propofol. Fentanyl is used for analgesia and atracurium is used for tracheal intubation.
  Interventions: Drug: Target controlled infusion of propofol; Drug: Fentanyl; Drug: Atracurium

INTERVENTIONS:
Device: bispectral index — Bispectral index (BIS) is one of several technologies used to monitor depth of anesthesia.
  Arms: bispectral index/TCI propofol/fentanyl
Drug: Target controlled infusion of propofol — TCI propofol (3-7 mcg/dL, Schnider model) is used for total intravenous anesthesia in both groups
  Other Names: TCI propofol
Drug: Fentanyl — Fentanyl 1-2 mcg/kg iv for induction and then 0.5-1.0 mcg/kg/hr infusion is used for analgesic.
Drug: Atracurium — Atracurium 0.6 mg/kg is used for endotracheal intubation
  Other Names: Tracrium

SUMMARY:
BIS is one of several equipments used to monitor depth of anesthesia.Some studies found BIS can reduce total propofol dose when being used with target controlled infusion (TCI).The objective is to compare awakening time after spine surgery between using clinical signs and bispectral index (BIS) guided target controlled infusion(TCI) of propofol in patients having neurophysiologic monitoring.

DETAILED DESCRIPTION:
34 patients undergoing spine surgery will be enrolled and randomly assigned into two groups. We exclude patients who age under 18 and over 80 years, preoperative hemodynamics instability, propofol allergy, receiving drugs interfered with EEG, liver disease, Body Mass Index (BMI) over 30 kg/m2. Before induction the patient will be given 0.9% Sodium Chloride (NaCl) or acetate Ringer solution 7 ml/kg. Standard monitorings are used to all patients.

Control group will receive fentanyl 1 mcg/kg and then fentanyl infusion 1 mcg/kg/hr and propofol TCI target 3-7 mcg/ml until asleep and then atracurium 0.5 mg/kg was given to facilitate endotracheal intubation. The patients will be ventilated with air:oxygen 1:1 L. The TCI propofol will be adjusted by clinical monitoring. If the patient has minor movement, the propofol TCI will be increased incrementally to 0.5 mcg/ml higher level but if major movement occurs the dose will be increased to1.0 mcg/ml higher. When hypotension occurs, this will be treated by fluid loading 200 ml in 10 min if it is not improved, then ephedrine or norepinephrine will be given and the TCI dose will be decreased by 0.5 mcg/ml lower level but not lower than 3.0 mcg/ml. Hypertension will be treated by fentanyl bolus 0.5 mcg/kg and increasing TCI dose to 0.5 mcg/ml higher level but not more than 7 mcg/ml. If hypertension persist, the nicardipine or diltiazem will be given.

Intervention group receives fentanyl 1 mcg/kg and then fentanyl infusion 1 mcg/kg/hr and propofol by TCI 3-7 mcg/ml until asleep and then atracurium 0.5 mg/kg was given to facilitate endotracheal intubation. The patients will be ventilated with air:oxygen 1:1 L. Propofol will be adjusted by BIS monitoring. If the movement occurs and BIS 40-60, fentanyl 0.5 mcg/kg will be given, BIS > 60, TCI dose will be increased 0.5 mcg/ml higher level until BIS 40-60. When hypotension occurs, if BIS 40-60, will be treated by load fluid 200 ml in 10 mins, then ephedrine or norepinephrine will be given, If BIS < 40 the TCI dose will decrease 0.5 mcg/ml but not lower than 3.0 mcg/ml. Hypertension occurs, if BIS > 60 will be treated by fentanyl bolus 0.5 mcg/kg and TCI dose will be increased 0.5 mcg/ml higher level but not more than 7 mcg/ml if not improved, nicardipine or diltiazem will be given. if BIS 40-60, nicardipine or diltiazem will be given.

This outcome measures are extubation time,total propofol dose.

ELIGIBILITY:
Inclusion Criteria:

* spine surgery with neurophysiology monitoring
* ASA 1-3
* elective case
* cooperate patients
* Not receive drugs interfere with EEG

Exclusion Criteria:

* unstable hemodynamics
* liver disease
* propofol allergy
* BMI > 30
* complete cord lesion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manee Raksakietisak, MD, Principal Investigator — Mahidol University
Locations (1):
- Mahidol University, siriraj hospital, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Bispectral Index: Bispectral index guides the target controlled infusion of propofol by keeping BIS 40-60 throughout operation.
- Clinical Signs: Clinical signs (heart rate, blood pressure and movement) guide target controlled infusion(TCI) of propofol.
Period: Overall Study
Arm/Group | Bispectral Index | Clinical Signs
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 40 patients met the inclusion criteria; however, three patients in each group were discontinued from the study due to protocol violation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bispectral Index | Clinical Signs | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.6) | 48.0 (12.1) | 49.05 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  Thailand | 17 | 17 | 34
Body weight [Mean (Standard Deviation); unit: kg] | 62.8 (11.8) | 60.4 (8.1) | 61.6 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Extubation Time
Description: Awakening time from finished operation to endotracheal extubation.
Time Frame: 4 hr
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Bispectral Index | Clinical Signs
Number analyzed (Participants) | 17 | 17
min | 16.3 (9.7) | 16.6 (8.9)

2. Secondary Outcome: Total Propofol Dosage
Description: total propofol dosage = propofol dose from start to end of the operation
Time Frame: From start anesthesia to finish operation
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Bispectral Index | Clinical Signs
Number analyzed (Participants) | 17 | 17
mg | 2,146 (742) | 2,340 (839)

ADVERSE EVENTS:
Time Frame: From start anesthesia to 24 hr after operation.
Description: The cardiovascular, respiratory, neurological or other complications during the intraoperative period are recorded.
Arm/Group | Bispectral Index | Clinical Signs
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes